CLINICAL TRIAL: NCT03662724
Title: Registry Study on Patient Characteristics, Biological Disease Profile and Clinical Course in the Treatment of Acute Myeloid Leukemia With Venetoclax: The Venetoclax Registry
Brief Title: Venetoclax Registry
Acronym: VENreg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 7972_BO_K_2018
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapsed/refractory adult acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Samples with DNA (either bone marrow or peripheral blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Venetoclax — Registry study observing clinical and biological characteristics of patients with acute myeloid leukemia who are treated with Venetoclax.
  Other Names: Venclyxto

SUMMARY:
Registry Study on Patient Characteristics, Biological Disease Profile and Clinical Course in the Treatment of Acute Myeloid Leukemia With Venetoclax

DETAILED DESCRIPTION:
The aim of this study is to document all patients with AML who are treated with the BCL2 inhibitor Venetoclax outside a clinical trial in all hospitals participating in this registry study in a standardised manner. Data is collected retrospectively and multi-centric. It is neither a therapy study nor is the therapy influenced by this study.

1. Systematic and uniform collection and documentation of all patients treated with the BCL2 inhibitor Venetoclax.
2. Collection and integrative analysis of clinical data of included patients.
3. Mutation analysis of available patient samples and correlation with clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

relapsed/refractory AML

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiens with relapsed/refractory AML including patients who received stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of Venetoclax treatment. | 4 months
  Overall response rate of Venetoclax treatment (complete remission, complete remission with incomplete regeneration, partial remission)

SECONDARY OUTCOMES:
Event-free survival during Venetoclax treatment | 5 years
  Event-free survival of patients with relapsed/refractory AML receiving Venetoclax
Relapse-free survival during Venetoclax treatment | 5 years
  Relapse-free survival of patients with relapsed/refractory AML receiving Venetoclax
Overall survival during Venetoclax treatment | 5 years
  Overall survival of patients with relapsed/refractory AML receiving Venetoclax

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heuser, MD, Principal Investigator — Hannover Medical School; Rabia Shahswar, MD, Principal Investigator — Hannover Medical School; Gernot Beutel, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Medical School Hannover, Hanover, Lower Saxony, Germany